CLINICAL TRIAL: NCT02864823
Title: Autologous Perichondrium Transplantation for Replacement of Stem Cells and Their Niche in the Treatment of Necrotizing Scleritis
Brief Title: Perichondrium Autograft in Refractory Necrotizing Scleritis
Acronym: PCRNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Collaborators: Ministry of Science and ICT, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jae Chan Kim, Professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRNS-1
Record Dates: First submitted 2016-07-21; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Necrotizing Scleritis
Keywords: Scleromalacia perforans; Necrotizing Scleritis; Perichondrium
MeSH Terms: conditions — Scleritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perichondrium (Experimental): Perichondrium Autografts
  Interventions: Procedure: Perichondrium Autografts

INTERVENTIONS:
Procedure: Perichondrium Autografts — Perichondrium tissue was harvested from the patient's ear cartilage and transplanted to reconstruct the scleral defect.
  Other Names: Perichondrium Transplantation

SUMMARY:
Necrotizing scleritis with severe ischemia is refractory to conventional treatment because of avascular necrosis.

The investigators assessed the therapeutic efficacy and safety of autologous perichondrium transplantation in patients with severe ischemic necrotizing scleritis, and analyzed the therapeutic effects.

DETAILED DESCRIPTION:
Ischemic necrotizing scleritis patients who showed persistent and progressive scleral melting were included in this study.

Perichondrium tissue was harvested from the patient's ear cartilage and transplanted to reconstruct the scleral defect after the necrotic tissue removal.

ELIGIBILITY:
Inclusion Criteria:

1. impending perforation or perforation state of sclera;
2. graft melting following previous surgery;
3. bacterial or fungal infection of sclera or graft after previous surgery;
4. discomfort due to protrusion of scleral calcification with ischemic necrosis
5. broad avascular area larger than 10 mm in diameter

Exclusion Criteria:

1. asymptomatic patients
2. smaller scleral defect less than 10 mm in diameter
3. shallow scleral defect

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Success Rate of Repair of Scleral Defects | Six months after reconstructive surgery
  Success Rate of Repair of Scleral Defects

SECONDARY OUTCOMES:
Post-Operative Complications | Six months after reconstructive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jae Chan Kim, Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Jee Taek Kim, Ph.D., Study Director — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung Ang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Watson PG, Hayreh SS, Awdry PN. Episcleritis and scleritis. I. Br J Ophthalmol. 1968 Mar;52(3):278-9 contd. doi: 10.1136/bjo.52.3.278. No abstract available. PMID 5650814
- [Background] Mamalis N, Johnson MD, Haines JM, Teske MP, Olson RJ. Corneal-scleral melt in association with cataract surgery and intraocular lenses: a report of four cases. J Cataract Refract Surg. 1990 Jan;16(1):108-15. doi: 10.1016/s0886-3350(13)80884-x. PMID 2299561
- [Background] Sainz de la Maza M, Foster CS, Jabbur NS. Scleritis associated with systemic vasculitic diseases. Ophthalmology. 1995 Apr;102(4):687-92. doi: 10.1016/s0161-6420(95)30970-0. PMID 7724185
- [Background] Torchia RT, Dunn RE, Pease PJ. Fascia lata grafting in scleromalacia perforans with lamellar corneal-scleral dissection. Am J Ophthalmol. 1968 Oct;66(4):705-9. doi: 10.1016/0002-9394(68)91293-2. No abstract available. PMID 5729586
- [Background] Yalcindag FN, Celik S, Ozdemir O. Repair of anterior staphyloma with dehydrated dura mater patch graft. Ophthalmic Surg Lasers Imaging. 2008 Jul-Aug;39(4):346-7. doi: 10.3928/15428877-20080701-19. PMID 18717447
- [Background] Breslin CW, Katz JI, Kaufman HE. Surgical management of necrotizing scleritis. Arch Ophthalmol. 1977 Nov;95(11):2038-40. doi: 10.1001/archopht.1977.04450110132017. PMID 921583
- [Background] Koenig SB, Kaufman HE. The treatment of necrotizing scleritis with an autogenous periosteal graft. Ophthalmic Surg. 1983 Dec;14(12):1029-32. PMID 6672701
- [Background] Ma DH, Wang SF, Su WY, Tsai RJ. Amniotic membrane graft for the management of scleral melting and corneal perforation in recalcitrant infectious scleral and corneoscleral ulcers. Cornea. 2002 Apr;21(3):275-83. doi: 10.1097/00003226-200204000-00008. PMID 11917176
- [Background] Sainz de la Maza M, Tauber J, Foster CS. Scleral grafting for necrotizing scleritis. Ophthalmology. 1989 Mar;96(3):306-10. doi: 10.1016/s0161-6420(89)32892-2. PMID 2710520
- [Background] Araf D, Moura Eda M, Rodrigues CJ, Figueiredo LA. [Homologous scleral and dura mater grafts in rabbit eyes: a comparative histopathological analysis]. Arq Bras Oftalmol. 2007 Nov-Dec;70(6):981-7. doi: 10.1590/s0004-27492007000600018. Portuguese. PMID 18235911
- [Background] Beaver HA, Patrinely JR, Holds JB, Soper MP. Periocular autografts in socket reconstruction. Ophthalmology. 1996 Sep;103(9):1498-502. doi: 10.1016/s0161-6420(96)30477-6. PMID 8841312
- [Background] Bairati A, Comazzi M, Gioria M. A comparative study of perichondrial tissue in mammalian cartilages. Tissue Cell. 1996 Aug;28(4):455-68. doi: 10.1016/s0040-8166(96)80031-0. PMID 8760859
- [Background] Togo T, Utani A, Naitoh M, Ohta M, Tsuji Y, Morikawa N, Nakamura M, Suzuki S. Identification of cartilage progenitor cells in the adult ear perichondrium: utilization for cartilage reconstruction. Lab Invest. 2006 May;86(5):445-57. doi: 10.1038/labinvest.3700409. PMID 16625212
- [Background] Casas VE, Kheirkhah A, Blanco G, Tseng SC. Surgical approach for scleral ischemia and melt. Cornea. 2008 Feb;27(2):196-201. doi: 10.1097/ICO.0b013e31815ba1ae. PMID 18216576
- [Background] Seko Y, Azuma N, Takahashi Y, Makino H, Morito T, Muneta T, Matsumoto K, Saito H, Sekiya I, Umezawa A. Human sclera maintains common characteristics with cartilage throughout evolution. PLoS One. 2008;3(11):e3709. doi: 10.1371/journal.pone.0003709. Epub 2008 Nov 12. PMID 19002264
- [Background] Franz-Odendaal TA, Vickaryous MK. Skeletal elements in the vertebrate eye and adnexa: morphological and developmental perspectives. Dev Dyn. 2006 May;235(5):1244-55. doi: 10.1002/dvdy.20718. PMID 16496288
- [Background] Koob TJ, Lim JJ, Massee M, Zabek N, Rennert R, Gurtner G, Li WW. Angiogenic properties of dehydrated human amnion/chorion allografts: therapeutic potential for soft tissue repair and regeneration. Vasc Cell. 2014 May 1;6:10. doi: 10.1186/2045-824X-6-10. eCollection 2014. PMID 24817999
- [Background] Smith JR, Mackensen F, Rosenbaum JT. Therapy insight: scleritis and its relationship to systemic autoimmune disease. Nat Clin Pract Rheumatol. 2007 Apr;3(4):219-26. doi: 10.1038/ncprheum0454. PMID 17396107
- [Background] Boccieri A, Marianetti TM. Perichondrium graft: harvesting and indications in nasal surgery. J Craniofac Surg. 2010 Jan;21(1):40-4. doi: 10.1097/SCS.0b013e3181c362df. PMID 20061978